CLINICAL TRIAL: NCT03975400
Title: Using Digital Media Advertising to Reduce the Duration of Untreated Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 19-0266; 5R34MH120790-03 (NIH)
Record Dates: First submitted 2019-05-30; First posted 2019-06-05 (Actual); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Schizophrenia; First Episode Psychosis
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Campaign (No Intervention): Investigators will measure the duration of untreated psychosis and rates of referrals to OnTrackNY programs throughout New York States prior to campaign initiation.
- Active Campaign (Active Comparator): Investigators will measure the duration of untreated psychosis and rates of referrals to OnTrackNY programs throughout New York States during the active campaign initiation.
  Interventions: Behavioral: search engine advertisement campaign

INTERVENTIONS:
Behavioral: search engine advertisement campaign — This proposal aims to explore whether targeted and proactive online outreach through search engine advertisements, coupled with engaging, informative, and interactive online resources, can effectively reduce the duration of untreated psychosis and facilitate earlier treatment initiation in New York State.
  Arms: Active Campaign

SUMMARY:
There is compelling evidence that longer duration of untreated psychosis independently predicts negative outcomes. The proposal aims to explore whether targeted and proactive online outreach through search engine advertisements, coupled with engaging, informative, and interactive online resources, can effectively reduce the duration of untreated psychosis and facilitate earlier treatment initiation in New York State. Results from this initiative will be critical to informing the subsequent design and conduct of larger, focused, and proactive digital media campaigns targeting patient with First Episode Psychosis and their caregivers online, intended to accelerate linkage to care and reduce the duration of untreated psychosis throughout the U.S.

DETAILED DESCRIPTION:
Approximately 100,000 individuals in the Unites States experience a first episode of psychosis (FEP) each year. Psychotic symptoms typically emerge during formative years of adolescence and young adult development and interfere with the establishment of healthy educational, vocational, and social foundations. Despite the severity of symptoms and significant decline in functioning, the time between symptom onset and receiving appropriate care in the U.S. is alarmingly lengthy. Longer Duration of Untreated Psychosis (DUP) has been shown to independently predict negative outcomes, including poorer response to treatment, worse global, vocational, social, and cognitive functioning, greater risk of relapse, higher symptom severity, and poorer quality of life. Prior successful DUP reduction initiatives have utilized various marketing strategies to educate the community about early intervention services, however these strategies are expensive, inefficient, and outdated. Targeted online outreach, supported by technological innovation, offers the prospect of proactively reaching individuals earlier in the course of illness development, as well as individuals who might not otherwise come into contact with traditional referral sources. In response to this challenge, Northwell Health's early psychosis research team is collaborating with Strong365, a nonprofit initiative dedicated to raising early psychosis intervention awareness, to develop and test a proactive and targeted comprehensive digital media marketing campaign designed to facilitate help-seeking and encourage treatment initiation in prospective patients with FEP and their caregivers. Investigators will take advantage of search engine advertisements, which allow advertisers (researchers) to select keywords/phrases and create linked ads appearing as a strategically placed search result. Dedicated ads will appear in response to online search queries conducted by prospective patients and their caregivers throughout New York State (NYS) that align with the campaign's pre-selected keywords/phrases. Individuals who click on the ads will be immediately directed to a landing page/website, and offered a variety of innovative and interactive online engagement tools intended to instantly connect users with specialty care staff and to facilitate earlier treatment initiation. Campaign referrals will be centralized and individuals with FEP will be enrolled into OnTrackNY (OTNY), a network of 21 dedicated early psychosis intervention programs throughout NYS. The campaign will target individuals as well as their caregivers, searching for psychosis-related terms or information online. Investigators will measure the DUP of individuals enrolled into OTNY before and after campaign activation and track the impact of the campaign on the number of FEP referrals and number of patients admitted to OTNY in NYS. Furthermore, investigators aim to identify the campaign target audience most effective at promoting treatment initiation as well as the online tools and resources most effective at encouraging treatment initiation for individuals with FEP. Investigators will additionally explore the online trajectories to care of individuals with FEP engaging with the campaign.

ELIGIBILITY:
Inclusion Criteria: All individuals searching online for information related to mental health

Exclusion Criteria: none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Birnbaum, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - Northwell, Glen Oaks, New York
  - Northwell, Queens, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A stepped-wedge cluster randomization design was implemented. OTNY sites were grouped into 6 clusters/regions based on geolocation and the total number of referrals received at each clinic. The six clusters/regions were; 1) Bronx, 2) Manhattan, 3) Queens, 4) Brooklyn, 5) Hudson River/Central NY, 6) Staten Island/Long-Island/Western NY. There was a total of four 6-month time periods, including the baseline period where all 6 clusters receive the control treatment.
Units Other Than Participants: Regions
Groups:
- Manhattan and Queens: 6 months control: 18 months campaign. After the initial 6-month baseline period, the campaign began running in 2 regions in NYS including Manhattan (4 sites) and Queens (3 sites). The campaign remained active for the entire 18 months.
  All other regions/sites remained in the control condition (no campaign).
- Brooklyn and Hudson Valley/Central NY/Westchester/Middleton: 12 months control; 12 months campaign. After 12 months in the control condition, the campaign expanded to another 2 regions including Brooklyn (3 sites), Hudson Valley/Central NY/Westchester/Middleton (6 sites).
  All other regions/sites remained in the control condition (no campaign).
- Bronx and Staten Island/Long Island/Western NY: 18 months control; 6 months active campaign. After 18 months in the control condition, the campaign expanded to the final 2 regions including the Bronx (2 sites) and Staten Island/Long Island/Western NY (4 sites).
Period: Baseline: Pre-Campaign Activation
Arm/Group | Manhattan and Queens | Brooklyn and Hudson Valley/Central NY/Westchester/Middleton | Bronx and Staten Island/Long Island/Western NY
Started (6-month baseline period where all regions were in the control condition (no campaign).) | 65; 2 Regions (Campaign activation period across NY state) | 84; 2 Regions | 42; 2 Regions
Completed | 65; 2 Regions | 84; 2 Regions | 42; 2 Regions
Not Completed | 0; 0 Regions | 0; 0 Regions | 0; 0 Regions
Period: Phase 1 (Active in 2 Regions)
Arm/Group | Manhattan and Queens | Brooklyn and Hudson Valley/Central NY/Westchester/Middleton | Bronx and Staten Island/Long Island/Western NY
Started (Campaign activated in Manhattan and Queens) | 62; 2 Regions | 79; 2 Regions | 42; 2 Regions
Completed | 62; 2 Regions | 79; 2 Regions | 42; 2 Regions
Not Completed | 0; 0 Regions | 0; 0 Regions | 0; 0 Regions
Period: Phase 2 (Active in 4 Regions)
Arm/Group | Manhattan and Queens | Brooklyn and Hudson Valley/Central NY/Westchester/Middleton | Bronx and Staten Island/Long Island/Western NY
Started (Campaign expanded to Brooklyn and Hudson Valley/Central NY/Westchester/Middleton) | 54; 2 Regions | 78; 2 Regions | 44; 2 Regions
Completed | 54; 2 Regions | 78; 2 Regions | 44; 2 Regions
Not Completed | 0; 0 Regions | 0; 0 Regions | 0; 0 Regions
Period: Phase 3 (Active in All 6 Regions)
Arm/Group | Manhattan and Queens | Brooklyn and Hudson Valley/Central NY/Westchester/Middleton | Bronx and Staten Island/Long Island/Western NY
Started (Campaign expanded to Bronx and Staten Island/Long Island/Western NY) | 55; 2 Regions | 52; 2 Regions | 41; 2 Regions
Completed | 55; 2 Regions | 52; 2 Regions | 41; 2 Regions
Not Completed | 0; 0 Regions | 0; 0 Regions | 0; 0 Regions

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Campaign | Active Campaign | Total
Number analyzed (Participants) | 356 | 342 | 698
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.03 (0.13) | 21.26 (0.21) | 21.17 (0.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 105 | 212
  Male | 249 | 237 | 486
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 80 | 57 | 137
  Not Hispanic or Latino | 238 | 227 | 465
  Unknown or Not Reported | 38 | 58 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 34 | 34 | 68
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 151 | 139 | 290
  White | 124 | 111 | 235
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 41 | 51 | 92

OUTCOME MEASURES:

1. Primary Outcome: Reducing the Duration of Untreated Psychosis
Description: Evaluate the effectiveness of a search engine ad campaign on reducing the duration of untreated psychosis (DUP) by directly comparing DUP pre-campaign to DUP during the campaign.
Time Frame: 2 years
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Pre-Campaign | Active Campaign
Number analyzed (Participants) | 356 | 342
Days | 5.32 (0.06) | 5.38 (0.09)

2. Secondary Outcome: Rates of Referrals
Description: Evaluate the effectiveness of a search engine ad campaign on rates of referrals by directly comparing referrals pre-campaign to referrals during the campaign.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: number of new referrals
Groups:
- Pre-Campaign: Investigators will measure the rates of referrals to OnTrackNY programs throughout New York States prior to campaign initiation.
- Active Campaign: Investigators will measure the rates of referrals to OnTrackNY programs throughout New York States during the active campaign initiation.
Arm/Group | Pre-Campaign | Active Campaign
Number analyzed (Participants) | 356 | 342
number of new referrals | 86.29 (26.10) | 32.10 (5.38)

ADVERSE EVENTS:
Time Frame: 2 years and 6 months
Description: Definition did not differ.
Arm/Group | Pre-Campaign | Active Campaign
All-Cause Mortality (participants affected / at risk) | 0/356 | 0/342
Serious Adverse Events (participants affected / at risk) | 0/356 | 0/342
Other Adverse Events (participants affected / at risk) | 0/356 | 0/342

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT03975400/Prot_SAP_000.pdf